CLINICAL TRIAL: NCT03338881
Title: A Phase 1 Study to Assess Mass Balance, Pharmacokinetics, and Metabolism of Orally Administered [14 C]-TAK-659 in Patients With Advanced Solid Tumor and/or Lymphoma Malignancies
Brief Title: A Study to Assess Mass Balance, Pharmacokinetics (PK), and Metabolism of Orally Administered [14 C]-TAK-659 in Participants With Advanced Solid Tumor and/or Lymphoma Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision: no safety or efficacy concerns
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C34010; U1111-1203-6940 (Other: World Health Organization); 2017-003383-12 (EudraCT Number)
Record Dates: First submitted 2017-11-08; First posted 2017-11-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Neoplasms; Lymphoma Neoplasms
Keywords: Drug therapy
MeSH Terms: interventions — TAK-659

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-TAK-659 100 mg (Experimental): [14C]-TAK-659 100 mg, solution, orally, once, in the fasted state on Day 1. Participant will have the option to continue treatment with TAK-659 100 mg, tablets, orally, once daily in a 28-day treatment cycle for up to 12 months or until disease progression or unacceptable toxicity, or the start of another anticancer therapy in post-ADME study period.
  Interventions: Drug: [14C]-TAK-659; Drug: TAK-659

INTERVENTIONS:
Drug: [14C]-TAK-659 — [14C]-TAK-659 solution.
Drug: TAK-659 — TAK-659 tablets.

SUMMARY:
The purpose of this study is to assess the mass balance and to characterize the pharmacokinetics (PK) in plasma and urine, and of total radioactivity in plasma and whole blood following a single oral dose of [14C]-TAK-659 solution containing 60 to 80 micro curie (Ci) of total radioactivity in participants with advanced solid tumors and/or lymphomas.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-659. TAK-659 is being tested to treat people who have advanced solid tumor and/or lymphoma malignancies. This study will look at the quantitative characterization of the mass balance, metabolic pathways, and rates and routes of excretion of TAK-659.

The study will enroll approximately 6 participants. The study will consist of 2 periods: absorption, distribution, metabolism, and excretion (ADME) study period and optional post-ADME study period. In ADME study period, participants will be assigned with [14C]-TAK-659 100 milligram (mg). After completion of ADME study period, participants may choose to continue in the optional post-ADME study period to receive TAK-659 100 mg.

This single center trial will be conducted in Netherlands. The overall time to participate in ADME study period will be 14 days and if participants choose the option to continue in the post-ADME study period, the maximum duration of participation will be 12 months, unless in the opinion of the investigator and sponsor the participant would derive benefit from continued treatment beyond 12 months. Participants will be followed up to 28 days after last dose of study drug or until the start of subsequent antineoplastic therapy, whichever occurs first.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have histologically or cytologically confirmed metastatic and/or advanced solid tumors and/or lymphomas for which standard curative or life-prolonging treatment does not exist or is no longer effective or tolerable.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
3. Life expectancy of at least 3 months.
4. Suitable venous access for the study-required blood sampling (that is, PK).
5. Recovered (that is, grade less than or equal to [<=] 1 toxicity) from the reversible effects of prior anticancer therapy (with the exception of alopecia and Grade 1 neuropathy).
6. Must have adequate organ function, including the following:

   * Adequate bone marrow reserve: absolute neutrophil count (ANC) greater than or equal to (>=) 1000 per microliter (/mcL); platelet count >=75,000/mcL (>=50,000/mcL for participants with bone marrow involvement); and hemoglobin >=8 gram per deciliter (g/dL) (red blood cell [RBC] and platelet transfusion allowed >=14 days before assessment).
   * Hepatic: total bilirubin <=1.5 times the upper limit of the normal range (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=2.5*ULN.
   * Renal: creatinine clearance >=60 milliliter per minute (mL/min) either as estimated by the Cockcroft-Gault equation or based on urine collection

Key Exclusion Criteria:

1. Central nervous system (CNS) lymphoma; active brain or leptomeningeal metastases, as indicated by positive cytology from lumbar puncture or computed tomography (CT) scan/magnetic resonance imaging (MRI).
2. Known human immunodeficiency virus (HIV) positivity or HIV-related malignancy.
3. Systemic anticancer treatment (including investigational agents) or radiotherapy within 3 weeks before the first dose of study treatment <=5 times the half-life for large molecule agents or <=4 weeks with evidence of progressive disease if 5 times the half-life is greater than (>) 4 weeks.
4. Use or consumption of any of the following substances:

   * Medications or supplements that are known to be inhibitors of P-glycoprotein (P-gp) and/or strong reversible inhibitors of cytochrome P450 (CYP) 3A within 5 times the inhibitor half-life (if a reasonable half-life estimate is known), or within 7 days (if a reasonable half-life estimate is unknown), before the first dose of study drugs
   * Medications or supplements that are known to be strong CYP3A mechanism-based inhibitors or strong CYP3A inducers and/or P-gp inducers within 7 days or within 5 times the inhibitor or inducer half-life (whichever is longer) before the first dose of study drugs. In general, the use of these agents is not permitted during the study except when an AE must be managed during interruption of study drug dosing.
   * Food or beverages containing grapefruit within 5 days before the first dose of study drugs. Note that food and beverages containing grapefruit are not permitted during the study.
5. Ongoing nausea or vomiting that is Grade 2 or worse in intensity.
6. Systemic infection requiring intravenous (IV) antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
7. Active secondary malignancy that requires treatment. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection and are considered disease-free at the time of study entry.
8. Irregular defecation patterns and/or history of urinary and/or fecal incontinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-10 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for TAK-659 | Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Cmax: Maximum Observed Plasma and Whole Blood Radioactivity for [14C]-TAK-659 | Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-659 | Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Tmax: Time to Reach the Maximum Plasma and Whole Blood Radioactivity for [14C]-TAK-659 | Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
AUClast: Area Under the Plasma Concentration-time Curve from Time 0 to the Time of the Last Quantifiable Concentration for TAK-659 | Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
AUClast: Area Under the Plasma and Whole Blood Radioactivity-time Curve from Time 0 to the Time of the Last Quantifiable Radioactivity for [14C]-TAK-659 | Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Ae urine,14C: Cumulative Amount of Radioactivity Excreted in Urine for [14C]-TAK-659 | Baseline up to 14 days
Ae feces, 14C: Cumulative Amount of Radioactivity Excreted in Feces for [14C]-TAK-659 | Baseline up to 14 days
Ae total: Total Cumulative Amount of Radioactivity Excreted in Urine and Feces for [14C]-TAK-659 | Baseline up to 14 days
Ae urine: Cumulative Amount of TAK-659 Excreted in Urine | Baseline up to 14 days
Percentage of Dose Excreted in Urine for TAK-659 | Baseline up to 14 days
Renal Clearance (CLR) of TAK-659 | Baseline up to 14 days

SECONDARY OUTCOMES:
Percentage of TAK-659 Metabolites in Plasma | Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Percentage of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline up to 28 days after the last dose of study drug (Week 58)
Percentage of Participants with Grade 3 or Higher Adverse Events (AEs) | Baseline up to 28 days after the last dose of study drug (Week 58)
Percentage of Participants with Drug Related AEs | Baseline up to 28 days after the last dose of study drug (Week 58)
Percentage of Participants with Drug Related Grade 3 or Higher AEs | Baseline up to 28 days after the last dose of study drug (Week 58)
Percentage of Participants with AEs Leading to Discontinuation of TAK-659 | Baseline up to 28 days after the last dose of study drug (Week 58)
Percentage of Participants who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose | Baseline up to 28 days after the last dose of study drug (Week 58)
Percentage of Participants who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose | Baseline up to 28 days after the last dose of study drug (Week 58)
Percentage of TAK-659 Metabolites in Urine and Feces | Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.